CLINICAL TRIAL: NCT01031628
Title: A Randomized, Phase 3 Study of Dose Escalation Versus No Dose Escalation of Imatinib In Metastatic GIST Patients With Imatinib Trough Levels Less Than 1100 Nanograms/mL
Brief Title: Study of Dose Escalation Versus no Dose Escalation of Imatinib in Metastatic Gastrointestinal Stromal Tumors (GIST) Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of feasibility secondary to slow accrual
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC019; STI571BUS286T
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Results first posted 2013-08-16 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST; Gastrointestinal stromal tumors; Exon 9; Gleevec; Imatinib blood levels
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (Active Comparator): Patients with blood level less than 1100 will continue imatinib 400 mg daily
  Interventions: Drug: Imatinib mesylate
- Arm B (Active Comparator): Patients with blood level less than 1100 dose adjust imatinib mesylate to goal blood level ≥1100 ng/mL
  Interventions: Drug: Imatinib mesylate
- Arm C (Active Comparator): Patients with blood level ≥1100 will continue imatinib 400 mg daily
  Interventions: Drug: Imatinib mesylate
- Arm D (Active Comparator): Patients with tumors that harbor exon 9 mutations will continue imatinib mesylate at 400 mg or dose escalate up to 800 mg daily
  Interventions: Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Imatinib mesylate — 400 mg daily. Number of cycles: until disease progression or unacceptable toxicity develops
  Other Names: Gleevec; Glivec
  Arms: Arm A; Arm C
Drug: Imatinib mesylate — 600 or 800 mg daily. Number of cycles: until disease progression or unacceptable toxicity develops
  Other Names: Gleevec; Glivec
  Arms: Arm B
Drug: Imatinib mesylate — 400, 600 or 800 mg daily. Number of cycles: until disease progression or unacceptable toxicity develops
  Other Names: Gleevec; Glivec
  Arms: Arm D

SUMMARY:
The purpose of this study is to determine if escalating the dose of imatinib to keep the drug blood level at ≥ 1100 ng/ml leads to better outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Unresectable and/or metastatic GIST
* Currently receiving imatinib 400 mg per day for a minimum of 4 weeks prior to registration, and for no more than 6 months prior to registration. This must be the first time that the patient has been treated for metastatic and/or unresectable GIST
* For patients who received imatinib following surgery at the time of an initial diagnosis of GIST, there must be a 6 month interval between completion of imatinib and the diagnosis of metastatic GIST
* Good physical functioning (ECOG Performance Status of 0 or 1)
* Generally, good function of organ such as liver and kidneys

Exclusion Criteria:

* Disease progression during adjuvant therapy with imatinib (adjuvant treatment is treatment that is given after surgery for GIST)
* Known intolerance of imatinib at a dose of 400 mg/day or higher
* Prior systemic therapy for advanced GIST with imatinib or those who have been on imatinib for longer than 6 months for unresectable and/or metastatic disease
* Major surgery within 2 weeks prior to Day 1 of study or who have not yet recovered from prior surgery
* Use of coumadin derivatives (i.e. warfarin, acenocoumarol, phenprocoumon)
* Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation < 2 weeks or who have not recovered from side effects of this therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne George, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (13):
- United States (13):
  - Cedars-Sinai Outpatient Cancer Center, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Carolinas Hematology Oncology Associates, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] George S, Trent JC. The role of imatinib plasma level testing in gastrointestinal stromal tumor. Cancer Chemother Pharmacol. 2011 Jan;67 Suppl 1:S45-50. doi: 10.1007/s00280-010-1527-2. Epub 2010 Dec 8. PMID 21140148
- [Derived] Marrari A, Trent JC, George S. Personalized cancer therapy for gastrointestinal stromal tumor: synergizing tumor genotyping with imatinib plasma levels. Curr Opin Oncol. 2010 Jul;22(4):336-41. doi: 10.1097/CCO.0b013e32833a6b8e. PMID 20489620
- See also: SARC Website — http://www.sarctrials.org

RESULTS

PARTICIPANT FLOW:
Groups:
- 400 mg for Patients With Imatinib Blood Levels < 1100: Patients with imatinib trough blood levels less than 1100 will continue imatinib 400 mg daily
  Imatinib mesylate : 400 mg daily. Number of cycles: until disease progression or unacceptable toxicity develops
- 600 or 800 mg for Patients With Imatinib Blood Levels < 1100: Patients with imatinib trough blood levels less than 1100 dose adjust imatinib mesylate to goal blood level ≥1100 ng/mL
  Imatinib mesylate : 600 or 800 mg daily. Number of cycles: until disease progression or unacceptable toxicity develops
- 400 mg for Patients With Imatinib Blood Levels ≥ 1100: Patients with imatinib trough blood levels ≥1100 will continue imatinib 400 mg daily
  Imatinib mesylate : 400 mg daily. Number of cycles: until disease progression or unacceptable toxicity develops
- 400, 600 or 800 mg for Patients With Exon 9 Mutation Tumors: Patients with tumors that harbor exon 9 mutations will continue imatinib mesylate at 400 mg or dose escalate up to 800 mg daily
  Imatinib mesylate : 400, 600 or 800 mg daily. Number of cycles: until disease progression or unacceptable toxicity develops
Period: Overall Study
Arm/Group | 400 mg for Patients With Imatinib Blood Levels < 1100 | 600 or 800 mg for Patients With Imatinib Blood Levels < 1100 | 400 mg for Patients With Imatinib Blood Levels ≥ 1100 | 400, 600 or 800 mg for Patients With Exon 9 Mutation Tumors
Started | 0 | 1 | 3 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 3 | 0
Not completed — Study terminated early | 0 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Patients with blood level less than 1100 will continue imatinib 400 mg daily
  Imatinib mesylate : 400 mg daily. Number of cycles: until disease progression or unacceptable toxicity develops
- Arm B: Patients with blood level less than 1100 dose adjust imatinib mesylate to goal blood level ≥1100 ng/mL
  Imatinib mesylate : 600 or 800 mg daily. Number of cycles: until disease progression or unacceptable toxicity develops
- Arm C: Patients with blood level ≥1100 will continue imatinib 400 mg daily
  Imatinib mesylate : 400 mg daily. Number of cycles: until disease progression or unacceptable toxicity develops
- Arm D: Patients with tumors that harbor exon 9 mutations will continue imatinib mesylate at 400 mg or dose escalate up to 800 mg daily
  Imatinib mesylate : 400, 600 or 800 mg daily. Number of cycles: until disease progression or unacceptable toxicity develops
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Total
Number analyzed (Participants) | 0 | 1 | 3 | 0 | 4
Age Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0 |  | 0
  Between 18 and 65 years |  | 0 | 3 |  | 3
  >=65 years |  | 1 | 0 |  | 1
Age Continuous [Mean (Standard Deviation); unit: years] |  | 71 | 56.7 (8.39) |  | 60.25 (7.68)
Gender [Number; unit: participants]
  Female |  | 1 | 1 |  | 2
  Male |  | 0 | 2 |  | 2
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 3 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Lesions for Progression or Response Via RECIST Criteria
Time Frame: Every 3 months
Population: Data were not collected or analyzed due to early termination.
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B | Arm C | Arm D
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1 | 2/3 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=0) | Arm B (N=1) | Arm C (N=3) | Arm D (N=0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysguesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
A decision was made to discontinue the SARC019 trial effective March 3, 2011, due to lack of feasibility secondary to slow accrual. Due to early termination of the study, no patients were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No